CLINICAL TRIAL: NCT04960306
Title: Fecal Filtrate Versus Conventional Microbiota Transplantation in the Treatment of Multiple Recurrent Clostridioides Difficile Infection (FILTRATE): A Protocol of a Randomized, Controlled Trial
Brief Title: Fecal Filtrate as a Treatment Option of Multiple Recurrent Clostridioides Difficile Infection
Acronym: FILTRATE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr Hegyi Péter, Principal Investigator, Director of the Centre for Translational Medicine at University of Pécs, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30700-5/2021/EÜIG
Record Dates: First submitted 2021-06-27; First posted 2021-07-13 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Clostridium Difficile Infection; Recurrent Clostridium Difficile Infection
Keywords: fecal microbiota transplantation; fecal filtrate; recurrent infection
MeSH Terms: conditions — Clostridium Infections; Reinfection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal filtrate transplantation (Active Comparator): Patients randomized to the fecal filtrate transplantation group
  Interventions: Biological: Fecal filtrate transplantation
- Conventional fecal microbiota transplantation (Active Comparator): Patients randomized to the conventional fecal microbiota transplantation group
  Interventions: Biological: Conventional fecal microbiota transplantation

INTERVENTIONS:
Biological: Fecal filtrate transplantation — Patients will receive 5-8 encapsulated lyophilized fecal filtrate transplantations in enterosolvent, size "0" capsules. Before intervention patients will receive proton pump inhibitors and prokinetics. After the preparation, the participants will be instructed to swallow the capsules one by one within 5 minutes with fluid to help to swallow the capsules.
  Arms: Fecal filtrate transplantation
Biological: Conventional fecal microbiota transplantation — Patients will receive 5-8 encapsulated lyophilized conventional fecal microbiota transplantations in enterosolvent, size "0" capsules. Before intervention patients will receive proton pump inhibitors and prokinetics. After the preparation, the participants will be instructed to swallow the capsules one by one within 5 minutes with fluid to help to swallow the capsules.
  Arms: Conventional fecal microbiota transplantation

SUMMARY:
Clostridioides difficile infection (CDI) is one of the most common hospital-acquired infectious diseases with a high mortality rate (6-30%). The treatment of CDI, especially the recurrent form of the disease is still considered a challenge. The FILTRATE randomized controlled trial aims to investigate the safety and efficacy of fecal filtrate transplantation in the treatment of recurrent CDI and compare it with conventional fecal microbiota transplantation (FMT).

DETAILED DESCRIPTION:
The treatment of recurrent CDI is still a burden on the healthcare system. FMT is highly effective for the treatment of recurrent CDI, resulting in the resolution of CDI up to 100% of the cases. FMT also has a good short-term safety profile, however long-term events like transfer of multiresistant bacteria and other living microorganism is still a major problem. On the other hand, the fecal filtrate contains only bacterial debris, proteins, and antimicrobial compounds and not intact microorganisms.

The FILTRATE trial is a multicenter, two-arm randomized controlled trial, and aims to compare the safety and efficacy of fecal filtrate transplantation to conventional fecal microbiota transplantation (FMT) in the treatment of recurrent CDI. Adult patients with multiple recurrent (>1) CDIs will be randomized 1:1 to receive either FMT or fecal filtrate transplantation. The transplantation will be carried out using lyophilized capsule on each arm. The primary endpoint of the study will be the clinical resolution of CDI-associated diarrhea 8 weeks after the interventions. Questionnaires will be completed on enrollment and at the time of each follow-up. Adverse events will be recorded and reported to the relevant institutional and national ethics committee. After the intervention, a one-year follow-up is also planned. Blood and stool samples will be collected at baseline and at each follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* multiple recurrent CDI (≥2 previous episodes of CDI)
* at least 3 or more loose or watery stools (Bristol 5-7) per day
* a positive Glutamate Dehydrogenase (GDH)-enzyme and positive CDI toxin A and/or B test
* the patient or the legal guardian sign the written informed consent

Exclusion Criteria:

* pregnancy or breastfeeding
* ongoing antibiotic treatment
* fulminant CDI
* previous FMT
* immunodeficiency
* need of intensive care
* requirement for vasoactive drugs
* other cause of diarrhea
* inflammatory bowel diseases
* irritable bowel syndrome
* life expectancy shorter than 3 months
* unavailable for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Resolution of diarrhea | 8 weeks
  Clinical resolution of the CDI associated diarrhea, defined by 2 or less stools (Bristol 1-4) per day in two consecutive days. The rate of the outcome will be compared within groups.

SECONDARY OUTCOMES:
Resolution of diarrhea | 1 year
  Clinical resolution of the CDI associated diarrhea, defined by 2 or less stools (Bristol 1-4) per day in two consecutive days. The rate of the outcome will be compared within groups.
Recurrence of CDI symptoms | 8 weeks, 1 year
  Recurrence of the CDI symptoms (diarrhea, abdominal pain ect.) within 8 weeks after an initial amelioration. The rate of the outcome will be compared within groups.
Overall mortality | 8 weeks, 1 year
  Overall mortality. The rate of the outcome will be compared within groups.
Disease associated mortality | 8 weeks, 1 year
  Disease-associated mortality. The rate of the outcome will be compared within groups.
Adverse events | 8 weeks, 1 year
  Proportion of adverse events (AE) and serious adverse events (SAE). The rate of the outcome will be compared within groups.
Change of the intestinal microbiome | 8 weeks, 1 year
  Change of the intestinal microbiome at the end of the follow up period regarding to the initial intestinal microbiome. The rate of the outcome will be compared within groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Translational Medicine, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Varga A, Kocsis B, Sipos D, Kasa P, Vigvari S, Pal S, Dembrovszky F, Farkas K, Peterfi Z. How to Apply FMT More Effectively, Conveniently and Flexible - A Comparison of FMT Methods. Front Cell Infect Microbiol. 2021 Jun 4;11:657320. doi: 10.3389/fcimb.2021.657320. eCollection 2021. PMID 34150673
- [Result] Dembrovszky F, Gede N, Szakacs Z, Hegyi P, Kiss S, Farkas N, Molnar Z, Imrei M, Dohos D, Peterfi Z. Fecal Microbiota Transplantation May Be the Best Option in Treating Multiple Clostridioides difficile Infection: A Network Meta-Analysis. Infect Dis Ther. 2021 Mar;10(1):201-211. doi: 10.1007/s40121-020-00356-9. Epub 2020 Oct 26. PMID 33106983
- [Result] Youngster I, Sauk J, Pindar C, Wilson RG, Kaplan JL, Smith MB, Alm EJ, Gevers D, Russell GH, Hohmann EL. Fecal microbiota transplant for relapsing Clostridium difficile infection using a frozen inoculum from unrelated donors: a randomized, open-label, controlled pilot study. Clin Infect Dis. 2014 Jun;58(11):1515-22. doi: 10.1093/cid/ciu135. Epub 2014 Apr 23. PMID 24762631
- See also: Related info — https://tm-centre.org/en/research/